CLINICAL TRIAL: NCT00648609
Title: Community Based Self Management of COPD Facilitated by a Palliative Care Team:Impact on Health Care Utilization and QOL
Status: Completed | Type: Observational
Sponsor: Essentia Health (Other)
Collaborators: Medica Sur Clinic & Foundation (Other)
Responsible Party: Dean Fox MD, St. Mary's Duluth Clinic Health System
Other Study IDs: 080801
Record Dates: First submitted 2008-03-27; First posted 2008-04-01 (Estimated); Last update posted 2011-06-20 (Estimated); Status verified 2011-06

CONDITIONS: Pulmonary Disease Chronic Obstructive
Keywords: Community based self management of COPD with palliative care
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Home-based palliative care services: Patients who are 60 or more years of age and have a diagnosis of COPD.Patients who have received two or more unscheduled acute care visits during the 12 months prior to the start of the study.
  Interventions: Other: Palliative home care in advanced COPD
- Standard of care: Patients who are 60 or more years of age and have a diagnosis of COPD.Patients who have received two or more unscheduled acute care visits during the 12 months prior to the start of the study.
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Palliative home care in advanced COPD — Interdisciplinary palliative care team on community based self care management of advanced COPD.
  Groups: Home-based palliative care services
Other: Standard of care — Usual care for COPD patients
  Groups: Standard of care

SUMMARY:
The purpose of this study is to compare in home support services for patients with COPD with usual care. The study is designed to evaluate the impact of an interdisciplinary palliative care team on community based self management of advanced COPD.

A total of thirty patients will be enrolled into this study. Twenty patients will be randomly assigned to receive usual care, and ten patients will be randomly assigned to usual care plus in home support services. This study will use objective criteria to identify patients with COPD likely to benefit from home based palliative care services. The patients will undergo initial assessment by medical, social work, and spiritual care personnel followed by a family meeting to establish a care plan. Periodic scheduled visits, and as needed unscheduled visits to address urgent needs will occur over one year's time in an attempt to return patients with COPD to the center of decision making regarding their care, avoid acute exacerbations and thereby avoid unscheduled clinic and ER visits. Patients will complete the QOL survey and symptom assessment scale upon initial intervention. After obtaining information from all patients who qualify for the study, participants will be randomized into cohorts. Those who are randomized to serve as cases will be provided with community based self management services by an interdisciplinary palliative care team. The control group will receive standard care. At the conclusion of 12 months both cases and controls will again complete the QOL survey,medical utilization, and symptom assessment.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 or greater
* Dx of COPD
* Received 2 or more unscheduled acute care visits during the 12 months from Jan 2007-Dec 2007
* SMDC primary care provider
* Lives within 50 miles of Duluth Minnesota
* Informed consent

Exclusion Criteria:

* Non English speaking
* Too ill or cognitively impaired to provide baseline data or informed consent
* Lives more than 50 miles from Duluth
* Nursing home resident

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced COPD from St. Mary's Duluth Clinic Health Systrem population in Duluth Minnesota
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2008-03; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Health service utilization, symptom scores, and patient quality of life | Baseline and 12 months
  Health care utilization: over 12 months while enrolled on study vs. 12 months prior to enrollment. For symptom scores and quality of life: at the time of enrollment and at the end of 12 months study period.

CONTACTS AND LOCATIONS:
Overall Officials: Dean Fox, MD, Principal Investigator — Essentia Health
Locations (1):
- Essentia Health, Duluth, Minnesota, United States

REFERENCES:
- [Background] Curtis JR, Engelberg RA, Wenrich MD, Au DH. Communication about palliative care for patients with chronic obstructive pulmonary disease. J Palliat Care. 2005 Autumn;21(3):157-64. PMID 16334970
- [Background] Halpern MT, Stanford RH, Borker R. The burden of COPD in the U.S.A.: results from the Confronting COPD survey. Respir Med. 2003 Mar;97 Suppl C:S81-9. doi: 10.1016/s0954-6111(03)80028-8. PMID 12647946
- [Background] Rocker GM, Sinuff T, Horton R, Hernandez P. Advanced chronic obstructive pulmonary disease: innovative approaches to palliation. J Palliat Med. 2007 Jun;10(3):783-97. doi: 10.1089/jpm.2007.9951. PMID 17592991
- [Background] American Academy of Hospice and Palliative Medicine; Center to Advance Palliative Care; Hospice and Palliative Nurses Association; Last Acts Partnership; National Hospice and Palliative Care Organization. National Consensus Project for Quality Palliative Care: Clinical Practice Guidelines for quality palliative care, executive summary. J Palliat Med. 2004 Oct;7(5):611-27. doi: 10.1089/jpm.2004.7.611. No abstract available. PMID 15588352
- [Background] Connors AF Jr, Dawson NV, Thomas C, Harrell FE Jr, Desbiens N, Fulkerson WJ, Kussin P, Bellamy P, Goldman L, Knaus WA. Outcomes following acute exacerbation of severe chronic obstructive lung disease. The SUPPORT investigators (Study to Understand Prognoses and Preferences for Outcomes and Risks of Treatments). Am J Respir Crit Care Med. 1996 Oct;154(4 Pt 1):959-67. doi: 10.1164/ajrccm.154.4.8887592.